CLINICAL TRIAL: NCT05764733
Title: The Bone, Exercise, Alendronate, and Caloric Restriction Trial
Brief Title: Bone, Exercise, Alendronate, and Caloric Restriction
Acronym: BEACON
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00077185; R01AG074979 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Bone Loss
Keywords: Older Adults; Weight Loss; Resistance Training; Osteoporosis; Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic; Weight Loss; Osteoporosis | interventions — Diphosphonates

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking applies to drug only. All assessments will be conducted by trained and blinded assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Resistance Training (RT) + Bisphosphonate (BIS) (Experimental): Progressive Resistance Training (RT) and Bone-Loading Exercise
  + 70 mg/weekly dose alendronate
  Interventions: Drug: Bisphosphonate; Behavioral: Resistance Training/Bone-Loading Exercise
- No RT + BIS (Experimental): No Resistance Training
  + 70 mg/weekly dose alendronate
  Interventions: Drug: Bisphosphonate
- No RT + Placebo (PL) (Active Comparator): No Resistance Training + Weekly Placebo
  Interventions: Other: Placebo
- RT + PL (Active Comparator): Progressive RT and Bone-Loading Exercise + Weekly Placebo
  Interventions: Behavioral: Resistance Training/Bone-Loading Exercise; Other: Placebo

INTERVENTIONS:
Drug: Bisphosphonate — Medicine used to treat bone problems, called osteopenia or osteoporosis.
  Arms: No RT + BIS; Resistance Training (RT) + Bisphosphonate (BIS)
Behavioral: Resistance Training/Bone-Loading Exercise — Exercise in small groups three days per week under the supervision of exercise physiologists. Heart rate and blood pressure will be measured before and after each session and participants will warm-up by walking or cycling for five minutes at a slow pace. All RT exercises will be conducted on machines which accommodate different body sizes and allow small increments in resistance, both important considerations for low functioning older adults with obesity.
  Arms: RT + PL; Resistance Training (RT) + Bisphosphonate (BIS)
Other: Placebo — Capsules identical to the active alendronate capsules without any active ingredients with the same dosing and follow up as BIS treatment group.
  Arms: No RT + Placebo (PL); RT + PL

SUMMARY:
The purpose of this research is to identify strategies that minimize bone loss that occurs when older adults lose weight. Participation in this research will involve up to nine assessment visits and last up to two years.

DETAILED DESCRIPTION:
The main objective of this study is to compare the independent and combined effects of a 12-month intervention of resistance training (RT) plus bone-loading exercises and bisphosphonate use on dietary weight loss (WL)-associated bone loss among older adults, with an indication for WL, and low bone density to explore lasting treatment efficacy. All participants will receive the same group-mediated dietary WL intervention and be randomized to one of four groups. Due to its robust change following dietary WL and clinical utility in predicting fracture, the study's primary outcome is change in total hip areal bone mineral density (aBMD) measured via dual x-ray absorptiometry (DXA). This will be complemented by DXA assessment at other skeletal sites, as well as high resolution peripheral quantitative computed tomography (HR-pQCT) derived compartmental volumetric (v)BMD, trabecular bone microarchitecture, cortical thickness/porosity, and strength at the distal radius and tibia allowing for assessment of intervention effectiveness on novel measures of bone quality.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* BMI>30 kg/m^2 or BMI 25.0 to <30 kg/m^2 plus one risk factor
* Currently receiving routine (annual) dental care
* Pre-existing low bone mass (T-score ≤-1.1 to >-2.5 at the hip, femoral neck, or lumbar spine (L1-L4))

Exclusion Criteria:

* Weight greater than 450 lbs (DXA limit)
* Resides with someone who is currently participating in BEACON
* Dependent on quad cane or walker; inability to walk independently
* History of mild cognitive impairment or dementia or evidence of cognitive impairment ((score <20) on Montreal Cognitive Assessment (MoCA))
* Excessive alcohol use (>21 drinks/week) in the past month; any non-cannabis illicit drug use
* Weight change ≥5% in past 3 months
* Regular participation (>60 mins per day on > 3 days/week) in structured strength training program for >6 months
* Severe arthritis, fracture, chronic injury, or other musculoskeletal disorder that prevents safe exercise participation; joint replacement or other orthopedic surgery in past 6 months or planned in next 12 months; invasive dental procedure (i.e. extraction/implant) in past 6 month or planned in next 12 months
* Osteoporosis (any of the following): Self-reported and on prescription osteoporosis medication; self-reported prior spine, hip, wrist, or shoulder fracture after age 40 (except when caused by trauma or fall from height), including atypical femoral fractures (AFF); or ≥20% for major osteoporotic fracture at screening
* Uncontrolled hypertension (systolic >180 OR diastolic >110 mmHg) upon repeated assessments (up to 3 times)
* Uncontrolled type 2 diabetes (HbA1c >8%); dialysis or abnormal kidney function (eGFR <45 mL/min/1.73 m2); liver disease or abnormal liver function (ALT levels 2 times above normal); anemia (Hb<LLN); calcium above or below normal limit; uncontrolled thyroid disease (hypo/hyper) or requiring recent (past 3 months) adjustments in thyroid hormone supplementation or thyroid-stimulating hormone <LLN or >10 mIU/ml; vitamin D deficiency (<20 ng/mL).
* Stroke, heart attack, heart failure hospitalization, or revascularization procedure within the past 6 months; chronic respiratory disease requiring oxygen; PAD diagnosis within the last 12 months; uncontrolled angina; progressive neurological disease; malabsorption disorder; any disease suggesting a life-expectancy <3 years; bilateral hip replacement; past or planned bariatric surgery; cancer requiring initial treatment within the last 12 months (except non-melanoma skin cancers); major vision or hearing loss; unstable gastric reflux; esophageal stricture, achalasia, or Barrett's esophagus
* Daily use of growth hormones, weight loss medications, oral steroids, or diabetes prescriptions (such as insulin, thiazolidinediones, or canagliflozin); known allergy to bisphosphonates; prior use of oral bisphosphonates for >3 months within the past 3 years; zoledronic acid within the past 5 years; denosumab use within the past year; anabolic agents for >3 months in the last year; current use of biotin or strontium; history of 3+ years of antiresorptive therapy
* Unable/unwilling to: provide own transportation to study visits, commit to study protocol (including random assignment), or adhere to data collection visits
* Current participation in another intervention research study; planned out-of-town trip greater than 1 month at a time during the first 6 months of the study; unwilling to provide informed consent, including consent to access personal electronic health records; judged unsuitable for the trial for any reason by research team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in total hip areal bone mineral density (aBMD) | from baseline through month 12
  Dual X-ray absorptiometry (DXA) derived

SECONDARY OUTCOMES:
aBMD assessment of the femoral neck | baseline, month 6, month 12
  DXA derived
aBMD assessment of the lumbar spine | baseline, month 6, month 12
  DXA derived
Tibial Trabecular (Tb) BMD | baseline and month 12
  HR-pQCT acquired; Average volumetric BMD [mg/cm3]
Tibial Cortical (Ct.) BMD | baseline, month 6, month 12
  HR-pQCT acquired; Avg. volumetric BMD [mg/cm3]
Tibial Trabecular Number (Tb.N) | baseline and month 12
  Average number trabeculae per unit length
Tibial Cortical Thickness (Ct.Th) | baseline and month 12
  Average thickness of cortical compartment in mm

OTHER OUTCOMES:
Tibial Total bone mineral density (Tt.BMD) | baseline and month 12
  High resolution peripheral quantitative computed tomography (HR-pQCT) acquired; Avg. volumetric BMD [mg/cm3]
Tibial Total Area (Tt.Ar) | baseline and month 12
  HR-pQCT acquired; Avg. cross-sectional area (all slices)
Tibial Trabecular Area (Tb Ar) | baseline and month 12
  HR-pQCT acquired; Avg. cross-sectional area (all slices)
Tibial Cortical Area (Ct.Ar) | baseline and month 12
  HR-pQCT acquired; Avg. cross-sectional area (all slices)
Tibial Total Trabecular Volume (Tt.TV) | baseline and month 12
  total Volume in tissue compartments; millimeter (mm)^3
Tibial Trabecular Volume (Tb.TV) | baseline and month 12
  Volumes in trabecular compartments; mm^3
Tibial Cortical Volume (Ct.TV) | baseline and month 12
  Volumes in cortical compartments; mm^3
Tibial Cortical Perimeter (Ct.Pm) | baseline and month 12
  millimeter; Average periosteal perimeter (all slices)
Tibial Trabecular Bone Volume Fraction (Tb.BV/TV) | baseline and month 12
  Volume ratio of bone in trabecular compartment percentage
Tibial Trabecular Thickness (Tb.Th) | baseline and month 12
  Average thickness of trabeculae in mm
Tibial Trabecular Separation (Tb.Sp) | baseline and month 12
  Avg distance between trabeculae in mm
Tibial Inhomogeneity of Trabecular Network | baseline and month 12
  Volume ratio of pores in cortical compartment
Tibial Cortical Porosity (Ct.Po) | baseline and month 12
  Volume ratio of pores in cortical compartment
Tibial Cortical Pore Diameter (Ct.Po.Dm) | baseline and month 12
  Average 3D diameter of pore volumes
Tibial Cortical Pore Volume (Ct.Po.V) | baseline and month 12
  Total volume of cortical pores
Tibial Estimated Failure Load (FL) | baseline and month 12
  Estimated by calculation of the reaction force at which 7.5% of the elements exceed a local effective strain of 0.7%
Tibial Bone Stiffness | baseline and month 12
  Reaction force divided by displacement
Bone Formation Assay | baseline, month 6, month 12
  Procollagen type I N-propeptide (PINP) is a biomarker of bone formation (mcg/L)
Bone Resorption Assay | baseline, month 6, month 12
  C-terminal telopeptide of type I collagen (CTX) is a biomarker of bone resorption (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Beavers, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beavers KM, Wolle BR, Ard JD, Beavers DP, Biehl O, Brubaker PH, Burghardt AJ, Calderone CT, Carballido-Gamio J, Fanning J, Kohrt WM, Love M, MacLean CM, Nicklas BJ, Stapleton J, Swanson CM, Weaver AA, Worden M, Wherry SJ. The Bone, Exercise, Alendronate, and Caloric Restriction (BEACON) trial design and methods. Contemp Clin Trials. 2024 Nov;146:107692. doi: 10.1016/j.cct.2024.107692. Epub 2024 Sep 17. PMID 39293778